CLINICAL TRIAL: NCT04672980
Title: A Phase 1 Study of RTX-321 for the Treatment of Patients With Advanced Malignancies Associated With Human Papillomavirus-16 Infection
Brief Title: RTX-321 Monotherapy in Patients With HPV 16+ Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The Sponsor terminated study after dosing 3 dose groups (9 pts) and closed trial on 11/30/22. RTX-321 was well-tolerated with no DLTs, no related deaths, SAEs or Gr. 3/4 AEs and cleared from circulation rapidly (w/in 10 min).
Sponsor: Rubius Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RTX-321-01
Record Dates: First submitted 2020-12-08; First posted 2020-12-17 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Cervical Cancer; Head and Neck Cancer; Anal Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Head and Neck Neoplasms; Anus Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RTX-321 Dose Escalation (Experimental): Phase 1: RTX-321 administered intravenously on Day 1 of each cycle monotherapy dose escalation
  Interventions: Drug: RTX-321
- RTX-321 Dose Expansion (Experimental): Phase 1: RTX-321 administered intravenously on Day 1 of each cycle.
  Interventions: Drug: RTX-321

INTERVENTIONS:
Drug: RTX-321 — RTX-321 monotherapy

SUMMARY:
This is an open-label, multicenter, multiple-ascending dose, FIH, Phase 1 study of RTX-321 for the treatment of patients that are HLA-A*02:01 positive with persistent, recurrent, or metastatic, unresectable, HPV 16+ cancers.

DETAILED DESCRIPTION:
This is a Phase 1, open label, multicenter, multidose, first-in-human (FIH) dose escalation and expansion to determine the safety and tolerability, recommended phase 2 dose and pharmacology, and antitumor activity of RTX-321 in adult patients with persistent, recurrent, or metastatic, unresectable cervical cancer (squamous, adeno, or adenosquamous histology), HNSCC, or squamous cell cancer of the anal canal that is not amenable to curative therapy. Prior to study screening, all patients must be confirmed to be HLA-A*02:01 positive. Documentation of an HPV 16+ tumor is required at prescreening for patients with cervical cancer and HNSCC. RTX-321 is a cellular therapy that expresses 4-1BBL, IL-12, and HPV-16 Antigen with the goal of harnessing the innate and adaptive immune systems for the treatment of cancer. The study will include a monotherapy dose escalation phase followed by an expansion phase.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent obtained prior to study procedures Patients ≥18 years with an ECOG 0 or 1
* Histologically confirmed diagnosis by the local laboratory of persistent, recurrent, or metastatic, unresectable cervical cancer (squamous, adeno, or adenosquamous histology), HNSCC, or squamous cell cancer of the anal canal that is not amenable to curative therapy.
* All patients must have experienced disease progression following platinum-based or mitomycin C-based chemotherapy administered in the persistent, recurrent, or metastatic setting.
* All patients with programmed death-ligand 1 (PD-L1) positive cervical cancer and those with HNSCC must have received or have been determined to be ineligible for immunotherapy with a PD-1 or PD-L1 inhibitor.
* All patients with cervical cancer will have received or have been determined to be ineligible for bevacizumab.
* Confirmation of HLA-A*02:01 positive status by central testing.
* In patients with cervical cancer or HNSCC, confirmation of HPV 16 within the tumor either from historical pathology result (using an FDA-approved HPV testing method, patients with cervical cancer only) or based on central laboratory analysis of a tumor sample. Patients with anal cancer will not be required to have prospective determination of HPV 16 positive status prior to enrollment.
* Disease must be measurable per Response Evaluation Criteria
* The shorter of 28 days or 5 half-lives must have elapsed since the completion of prior therapy, before initiation of study treatment.
* Adequate Organ Function as Defined by the protocol:

  * AST and ALT ≤3 × the upper limit of normal (ULN)
  * Except in documented cases of Gilbert syndrome, total bilirubin ≤1.5 × ULN
  * Serum albumin ≥2.5 g/dL
  * Serum or plasma creatinine ≤1.5 × ULN and/or glomerular filtration rate ≥50 mL/min/1.73 calculated by the Cockcroft-Gault formula
  * Absolute neutrophil count ≥1 × 103/μL, without myeloid growth factor support for ≥1 week
  * Platelet count ≥100 × 103/μL, without platelet transfusion for ≥1 week
  * Hemoglobin ≥9 g/dL, without red blood cell transfusion for ≥2 weeks

Exclusion Criteria:

* Patient has central nervous system (CNS) involvement. If the patient fulfills the following 3 criteria, she/he is eligible for the trial after consultation with the Sponsor Medical Monitor.

  * Completed prior therapy for CNS metastases (radiation and/or surgery)
  * CNS tumor(s) is clinically stable at the time of enrollment
  * Patient does not require corticosteroid or antiepileptic therapy for management of CNS metastases
* Known hypersensitivity to any component of study treatment or excipients.
* Positive antibody screen using institution's standard type and screen test.
* Clinically significant, active and uncontrolled infection, including human immunodeficiency virus (HIV), Hepatitis B virus (HBV), or Hepatitis C virus (HCV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Safety Assessment by rate of Adverse Events: | up to 30 months
  Measured by incidence of Treatment Emergent Adverse Events (TEAEs)
Dose limiting toxicities (DLTs) of RTX-321: | up to 30 months
  As determined by incidence and severity of adverse events (AEs)

SECONDARY OUTCOMES:
Pharmacodynamics (PD) of RTX-321: | up to 30 months
  As measured by the changes in number of CD8+ T-cells in peripheral blood using flow cytometry
Pharmacokinetics (PK) of RTX-321: | up to 30 months
  As measured by the detection of the number of RTX-321 cells using flow cytometry
Anti-tumor activity of RTX-321 | up to 30 months
  measured by duration of response (DoR)
Anti-tumor activity of RTX-321 | up to 30 months
  Measured by overall survival (OS)
Anti-tumor activity of RTX-321 | up to 30 months
  Measured by progression free survival (PFS)
Anti-tumor activity of RTX-321 | up to 30 months
  Measured by overall response rate (ORR)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - University of Alabama, Birmingham, Alabama
  - The Angeles Clinic & Research Institute, Los Angeles, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Washington University, St Louis, Missouri
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Virginia Cancer Specialists, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No